CLINICAL TRIAL: NCT03218020
Title: Red Meat Consumption and Risk of Cardiovascular Diseases - is Increased Iron Load a Possible Link?
Brief Title: Red Meat, Increased Iron Load and CVD Risk
Status: Completed | Type: Observational
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: DKFZ Study_ID 905
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Myocardial Infarction; Stroke; Cardiovascular Mortality
MeSH Terms: conditions — Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples from baseline examinations stored in the biobank of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Random Subcohort: Random subcohort (~10 % of the initial cohort, study has a case-cohort design; details on the case-cohort design have been described by Kulathinal et al., Epidemiol Perspect Innov, 2007: www.ncbi.nlm.nih.gov/pmc/articles/PMC2216006/).
  Interventions: Other: No intervention assigned, this is an observational study.
- Incident CVD Cases: Validated incident cases of myocardial infarction, stroke and CVD death that occured until Dec-31-2009 (details on the case-cohort design have been described by Kulathinal et al., Epidemiol Perspect Innov, 2007: www.ncbi.nlm.nih.gov/pmc/articles/PMC2216006/).
  Interventions: Other: No intervention assigned, this is an observational study.

INTERVENTIONS:
Other: No intervention assigned, this is an observational study. — No intervention assigned, this is an observational study.

SUMMARY:
Increased iron load could be a risk factor for cardiovascular diseases (CVD). Red meat consumption affects iron status and has also been shown to be related to increased CVD risk. The investigators hypothesized that risk associations between red meat intake and cardiovascular disease risk can to some degree be explained by higher iron load among individuals with higher meat intake. Thus, the investigators evaluate associations between red meat consumption, iron status, and CVD risk in a large-scale population based study, the European Prospective Investigation into Cancer and Nutrition (EPIC) - Heidelberg.

DETAILED DESCRIPTION:
The present study part of the the European Prospective Investigation into Cancer and Nutrition (EPIC) - Heidelberg, a large-scale observational cohort study located at the German Cancer Research Center, Heidelberg, Germany. The study started between 1994 and 1998, when 25 540 adults from the local general population were recruited. Study participants are being followed-up by active and passive procedures. The main aim of the study is to evaluate associations between diet, lifestyle as well as metabolism and risks of major chronic diseases (cancer, cardiovascular diseases, diabetes).

Here, the investigators register a project from within EPIC-Heidelberg on prediagnostic iron status as a potential mediator of associations between pre-diagnostic red meat consumption and cardiovascular disease risk. For this particular project, an embedded case-cohort set-up was chosen, i.e. iron status markers (primary marker: serum ferritin; secondary markers: serum transferrin, serum iron) were measured in baseline blood samples from a random subcohort (n=2738) and all validated incident cases of myocardial infarction (n=556), stroke (n=513), and CVD death (n=327) that occured until the closure date of the present study (12-31-2009).

Statistical analyses follow four steps to assess whether iron status may mediate associations between red meat consumption and CVD risk, as proposed by Wittenbecher et al. (Am J Clin Nutr, 2015: www.ncbi.nlm.nih.gov/pubmed/25948672):

1. Multivariable Cox regression analyses on red meat consumption and CVD risk, assuming a significant positive association
2. Multivariable linear regression analyses on red meat consumption and iron status, assuming a significant positive association
3. Multivariable Cox regression analyses on iron status and CVD risk, assuming a significant positive association
4. Multivariable Cox regression analyses on red meat consumption and CVD risk, additionally adjusting for iron status, assuming that the association will be attenuated by adjustment for iron status

ELIGIBILITY:
Inclusion Criteria:

General population, age 35-65 years

Exclusion Criteria:

Prevalent myocardial infraction or stroke

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: EPIC-Heidelberg was launched as part of EPIC-Europe between 1994 and 1998, when 13 611 female and 11 929 male participants aged 35 to 65 years were recruited from the local general population.
Sampling Method: Probability Sample
Enrollment: 25540 (Actual)
Dates: Start 1994-09-01 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Myocardial infraction | 1994 - 2009
  Incident cases of primary myocardial infarction according to clinical records
Stroke | 1994 - 2009
  Incident cases of primary stroke according to clinical records
Cardiovascular death | 1994 - 2009
  Incident cases of cardiovascular death according to death certificates

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Kaaks, Prof., Principal Investigator — German Cancer Research Center
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No